CLINICAL TRIAL: NCT00688311
Title: Pilot Trial of a Synbiotic in HIV+ Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: J William Critchfield/Associate Project Scientist, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 200715524-1
Record Dates: First submitted 2008-05-16; First posted 2008-06-02 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infection
Keywords: HIV; synbiotic; probiotic; immune activation; blood CD4 count; bacterial translocation; Human Immunodeficiency Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotic (Experimental): Ingestion of synbiotic dietary supplement
  Interventions: Dietary Supplement: Synbiotic 2000
- Placebo (Placebo Comparator): Ingestion of the Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic 2000 — A preparation consisting of 4 species of probiotic bacteria (10^10 each) combined with 4 types of dietary fiber (2.5g each).
  Other Names: Synbiotic 2000, Medipharm, Kagerod, Sweden
  Arms: Synbiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to test the hypothesis that daily ingestion of a 'synbiotic' for 4 weeks will improve intestinal function, ease immune system overactivation, and increase blood CD4 count in HIV-infected individuals. A 'Synbiotic' is a mixture of probiotic bacteria and dietary fiber.

DETAILED DESCRIPTION:
RATIONALE. HIV infection results in alterations to the intestinal tract, even in clinically healthy patients. Changes may include pronounced CD4 T-cell loss, enteric nerve and smooth muscle degeneration, abnormal enterocyte morphology, altered gene expression patterns, increased intestinal permeability, and decreased absorptive capacity. Recently it was found that HIV infection may also result in abnormal low-level leakage of lipopolysaccharide (LPS, a gram-negative bacterial product) from the gut into the circulation which promotes systemic immune activation. As immune activation is a strong positive correlate of HIV disease progression, it may be very important to develop effective means to improve intestinal barrier function in HIV infection. Evidence also exists that uninfected individuals of African descent may have higher intestinal permeability than uninfected Caucasians, suggesting that intestinal dysfunction in the event of HIV infection could differ between the two races. With regard to gender, women have been shown to display more pronounced inflammatory responses to LPS compared to men. Intriguing research outside the HIV field using animal models of compromised gut barrier function and also using human subjects with trauma- or disease-associated intestinal leakage has shown that oral administration of certain probiotic bacteria can 1) Reduce bacterial translocation, 2) Reduce bacterial infections, 3) Decrease inflammatory cytokines, and 4) Improve survival. Thus, probiotics could offer important benefits to HIV infected patients by improving intestinal function and reducing subsequent microbial translocation and immune activation. These benefits may vary by race.

OBJECTIVE. To determine the effect of an oral synbiotic supplement (Synbiotic 2000) on plasma LPS levels, systemic immune activation, and blood CD4 count in HIV infected women.

HYPOTHESIS. Oral treatment of HIV+ patients with this synbiotic supplement will improve intestinal barrier function, decrease the translocation of LPS into the circulation, and result in reduced systemic immune activation and improved CD4 count.

EXPERIMENTAL DESIGN. 30 HIV+ female subjects will be randomized to test supplement or placebo and undergo a baseline blood draw to establish initial values for plasma LPS, immune activation markers, and blood CD4 count. Following daily ingestion of the test supplement or placebo for 4 weeks, subjects will undergo a second blood draw for measurement of the same factors. Subjects will also provide a stool specimen at the beginning and end of the 4 week period.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Adult Female
* Currently taking antiretroviral medication

Exclusion Criteria:

* AIDS-defining conditions
* Current use of oral antibiotics
* Inflammatory bowel disease or other known GI pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Plasma Lipopolysaccharide | 4 weeks

SECONDARY OUTCOMES:
Immune Activation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bill Critchfield, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- CARES Clinic, Sacramento, California, United States

REFERENCES:
- [Background] Brenchley JM, Price DA, Schacker TW, Asher TE, Silvestri G, Rao S, Kazzaz Z, Bornstein E, Lambotte O, Altmann D, Blazar BR, Rodriguez B, Teixeira-Johnson L, Landay A, Martin JN, Hecht FM, Picker LJ, Lederman MM, Deeks SG, Douek DC. Microbial translocation is a cause of systemic immune activation in chronic HIV infection. Nat Med. 2006 Dec;12(12):1365-71. doi: 10.1038/nm1511. Epub 2006 Nov 19. PMID 17115046
- [Background] Rayes N, Seehofer D, Theruvath T, Schiller RA, Langrehr JM, Jonas S, Bengmark S, Neuhaus P. Supply of pre- and probiotics reduces bacterial infection rates after liver transplantation--a randomized, double-blind trial. Am J Transplant. 2005 Jan;5(1):125-30. doi: 10.1111/j.1600-6143.2004.00649.x. PMID 15636620
- [Background] Kotzampassi K, Giamarellos-Bourboulis EJ, Voudouris A, Kazamias P, Eleftheriadis E. Benefits of a synbiotic formula (Synbiotic 2000Forte) in critically Ill trauma patients: early results of a randomized controlled trial. World J Surg. 2006 Oct;30(10):1848-55. doi: 10.1007/s00268-005-0653-1. PMID 16983476
- [Background] Rayes N, Seehofer D, Theruvath T, Mogl M, Langrehr JM, Nussler NC, Bengmark S, Neuhaus P. Effect of enteral nutrition and synbiotics on bacterial infection rates after pylorus-preserving pancreatoduodenectomy: a randomized, double-blind trial. Ann Surg. 2007 Jul;246(1):36-41. doi: 10.1097/01.sla.0000259442.78947.19. PMID 17592288
- [Derived] Schunter M, Chu H, Hayes TL, McConnell D, Crawford SS, Luciw PA, Bengmark S, Asmuth DM, Brown J, Bevins CL, Shacklett BL, Critchfield JW. Randomized pilot trial of a synbiotic dietary supplement in chronic HIV-1 infection. BMC Complement Altern Med. 2012 Jun 29;12:84. doi: 10.1186/1472-6882-12-84. PMID 22747752